CLINICAL TRIAL: NCT02026843
Title: Analysis of Biomarkers From Patients With Chorioretinal Diseases
Status: Recruiting | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Park, Department of Opthalmology, School of medicine, Kyungpook National University, Kyungpook National University Hospital
Other Study IDs: KNUH2013-1
Record Dates: First submitted 2013-12-29; First posted 2014-01-03 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy; Macular Degeneration
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — certain gene or protein levels in ocular fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chorioretinal diseases: chorioretinal diseases including diabetic retinopathy, retinal vascular diseases, age-related macular degeneration (dry and wet), and retinal degeneration.
  Interventions: Drug: Chorioretinal diseases
- Control: control patients with surgeries include pars plana vitrectomy of macular hole, epiretinal membrane, cataract surgery.

INTERVENTIONS:
Drug: Chorioretinal diseases — chorioretinal diseases including diabetic retinopathy, retinal vascular diseases, age-related macular degeneration (dry and wet), and retinal degeneration
  Groups: Chorioretinal diseases

SUMMARY:
This study was conducted to investigate the levels of ocular biomarkers from the patients with chorioretinal diseases including diabetic retinopathy, retinal vascular diseases, age-related macular degeneration (dry and wet), and retinal degeneration.

DETAILED DESCRIPTION:
This prospective, case-control study included 50 patients(50eyes) with chorioretinal diseases including diabetic retinopathy, retinal vascular diseases, age-related macular degeneration (dry and wet), and retinal degeneration. and 50 patient with nondiabetic retinopathy or cataract. Ocular fluids and blood samples were taken before injection of anti-vascular endothelial growth factor agent or pars plana vitrectomy for other retinal disease. Ocular biomarkers were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age over 20 years
* patients requiring ophthalmologic treatments for different degrees of decreasing of visual acuity.
* patients with chorioretinal diseases including diabetic retinopathy, retinal vascular diseases, age-related macular degeneration (dry and wet), and retinal degeneration.
* control patients asking cataract surgery or vitrectomy for posterior segment nonproliferative disorders.

Exclusion Criteria:

* under the age of 20 years
* patients that received any anti-vascular endothelial growth factor agent for proliferative disease before taking sample of aqueous humor
* patients that did not signed the informed consent of the trial
* patients with intraocular inflammations or infections that requiring any pharmaceutical agent
* patients with recent ocular trauma

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients will be included. 50 patients with chorioretinal diseases including diabetic retinopathy, retinal vascular diseases, age-related macular degeneration (dry and wet), and retinal degeneration. and 50 control patients scheduled for pars plana vitrectomy for nondiabetic retinal disease or phacoemulsification.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2028-02 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Biomarkers in ocular fluids | one month
  To establish if certain type of chorioretinal diseases group are associated to different concentrations of gene or protein concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Park, M.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Dong Ho Park, Daegu, Kyungsangpookdo, South Korea

IPD SHARING:
Plan to Share IPD: No